CLINICAL TRIAL: NCT03783273
Title: The Influence of Food Matrix Delivery System on the Bioavailability of Vitamin D3
Acronym: DFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1107213017
Record Dates: First submitted 2018-12-07; First posted 2018-12-21 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-02

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D Insufficiency; Vitamin D Supplementation; Food Fortification
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Water; Milk

STUDY DESIGN:
Intervention Model Description: A multiple crossover study using a balanced latin square design. Each participant will receive all five treatments with a wash-out period of 10-21 days between each treatment.
Who Masked: Participant
Masking Description: Participants will not know if they receive juice with complex-bound vitamin D3 or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Whey protein complex-bound D3 + juice (Experimental): 200 microgram vitamin D3 in a whey protein-complex added to 500 mL of juice.
  Interventions: Dietary Supplement: Vitamin D3; Combination Product: Whey protein-complex; Other: Juice
- D3 + juice (Active Comparator): 200 microgram vitamin D3 added to 500 mL of juice.
  Interventions: Dietary Supplement: Vitamin D3; Other: Juice
- D3 + milk (Active Comparator): 200 microgram vitamin D3 added to 500 mL of skimmed-milk.
  Interventions: Dietary Supplement: Vitamin D3; Other: Milk
- D3 droplets (Active Comparator): 200 microgram vitamin D3 as droplets + 500 mL of water.
  Interventions: Dietary Supplement: Vitamin D3; Other: Water
- No vitamin D (Placebo Comparator): 500 mL of Water.
  Interventions: Other: Water

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Single dose vitamin D3
  Arms: D3 + juice; D3 + milk; D3 droplets; Whey protein complex-bound D3 + juice
Combination Product: Whey protein-complex — Whey protein complex-bound vitamin D3
  Arms: Whey protein complex-bound D3 + juice
Other: Water — 500 mL water
  Arms: D3 droplets; No vitamin D
Other: Milk — 500 mL milk
  Arms: D3 + milk
Other: Juice — 500 mL juice
  Arms: D3 + juice; Whey protein complex-bound D3 + juice

SUMMARY:
This study investigates the influence of different food matrices on the bioavailability of vitamin D.

Although most vitamin D comes from skin synthesis in response to sun exposure, dietary intake is also important - especially during winter time where there is no endogenous production of vitamin D in Denmark. A way to maintain an adequate vitamin D status is to supplement either as tablets/droplets or as fortified food. However, there seems to be an inter-individual variation in response to supplementation.

This study aims to investigate whether this variation in absorption of vitamin D may depend on delivery system.

DETAILED DESCRIPTION:
BACKGROUND The current project is a part of the vitamin D fortification with enhanced bioavailability study program (acronym: DFORT) which is an interdisciplinary project including research groups from Denmark, Spain, and the Netherlands supported by the Danish Innovation Foundation. The overall aim of DFORT is to develop more efficient strategies for vitamin D fortification by studying the influence of the delivery matrix on the bioavailability of vitamin D. DFORT is organized into four scientific work packages (WP).

The first two WPs have aimed to study whether complex formation (nano-encapsulation) of vitamin D with different proteins may enhance the stability of vitamin D (WP 1 lead by prof. Daniel Otzen, AU-iNANO) and the effect of complex formation in real food systems including investigations on the stability during storage, light- and heat-exposure (WP 2 lead by associate professor Trine Kastrup Dalsgaard, AU-FOOD). WP 1+2 have shown that vitamin D can be stabilized by complex formation with whey protein and that the encapsulation may cause less oxidative degradation thereby improving the stability of vitamin D in different food systems.

In the current study (WP 3 lead by prof. Lars Rejnmark, AU-Health), the bioavailability of vitamin D in different food matrices (including complex formation with whey protein) will be studied in humans. Biological samples will be collected in WP 3 allowing for metabolomics studies on possible associations between vitamin D supplementation through different food matrices and metabolic phenotype (WP 4 lead by prof. Hanne C. Bertram, AU-FOOD).

Although most of the total body vitamin D is synthesized in the skin after exposure to UV light (wavelength of 290-315 nm), most individuals require at least some dietary vitamin D to maintain a replete vitamin D status. This is especially true during wintertime. With a latitude of 56°N in Denmark, there is no endogenous synthesis of vitamin D in the months extending from October to April, which means that the inhabitants have to rely on food sources in order to maintain a replete vitamin D status. Cholecalciferol (vitamin D3 [D3]) is the main dietary source of vitamin D, but it is only present in a limited number of food items (such as fatty fish) making it difficult to achieve the recommended intake of 10 µg D3 per day.

Vitamin D status may be improved in response to an increased intake of vitamin D in terms of either supplementation with tablets or food fortification. Numerous studies have shown increased 25-hydroxy vitamin D (25OHD) levels in response to an increased intake of vitamin D. It is generally assumed that mean 25OHD concentrations increase by 0.7 nmol/L in response to an increased long-term intake of 1 µg vitamin D per day although the relative increase per microgram supplemented may be higher if baseline levels are low. Despite this well-known dose-response relationship in groups of people, several studies have documented that the change in serum 25OHD levels in response to vitamin D supplementation varies widely.

Several reasons may account for the inter-individual variation in response to vitamin D supplementation. In gross terms, the variation may be due to dosing inaccuracies (inconsistencies between claimed and actual values of vitamin D) and variation in bioavailability of vitamin D.

Inconsistencies between claimed and measured values of vitamin D content in vitamin D tablets and food-fortified products may be due to inconsistencies in dose used for fortification or to the instability of the vitamin per se. Discrepant results have been reported on the stability of vitamin D in different food matrices and when exposed to different physiochemical hazards. Some investigators have reported vitamin D to be unstable whereas others have found it to be remarkable stable when exposed to oxidation, light, and to acid and alkali.

Only few studies have searched for factors responsible for the inter-individual variation in 25OHD levels in response to vitamin D supplementation. These studies have suggested that body composition (including fat mass content), genetic variants of the vitamin D binding protein (VDBP), and the ratio of serum 24,25-dihydroxy vitamin D (24,25(OH)2D) to 25OHD may contribute to variation in serum 25OHD levels. However, in a recent study only 47% of the variations in the response to vitamin D supplementation could be explained by accounting for factors of known importance to changes in 25OHD levels.

In addition to the above-mentioned indices, factors of importance to the intestinal absorption of vitamin D as well as the food matrix by which vitamin D supplementation is provided may contribute to inter-individual variations in 25OHD responses. However, only few studies are available on the bioavailability of vitamin D from different food matrices and the intestinal absorption of vitamin D, including the intraluminal fate, and molecular mechanisms facilitating the absorption are still only partially understood.

As vitamin D is a fat-soluble molecule, it has generally been assumed that vitamin D is absorbed in the small intestine by simple passive diffusion with vitamin D being incorporated into the micelle and transported by chylomicrons via lymph veins to the liver. This is in alignment with studies showing an increased risk of low 25OHD levels in patients with fat malabsorption. Accordingly, it has been suggested that ingestion of vitamin D with a meal rich in fat may increase the release of bile, allowing an increased incorporation of vitamin D in the bile salt micelle thereby improving the bioavailability of vitamin D. However, discrepant results have been reported, on whether the composition of the food matrices (and its fat content) by which vitamin D is ingested influence its bioavailability.

In a randomized, controlled trial by Raimundo et al., the mean change in 25OHD levels two weeks after the treatment with a single large oral dose of 50,000 IU D3 was larger, when the meal had at least 15 g of fat compared to a fat-free meal. In contrast, the fat content of the food matrices was not found to influence the time-concentration profile as measured by vitamin D2 levels in plasma 2, 4, 8, 12, 48, and 72 h after ingestion of a single dose of 25,000 IU D2 added to either whole milk, skim milk or dissolved in 0.1 mL corn oil and applied to toast. However, both of these studies are limited by the use of very high (pharmacological) doses of vitamin D, which may override any physiological effects of the composition of the food matrices.

A lack of an effect of the fat content of the food by which vitamin D is ingested is also supported by studies on vitamin D fortification of orange juice. Comparing the bioavailability of vitamin D added to orange juice or supplemented as capsules showed a similar increase in 25OHD concentrations in response to 11 weeks of supplementation with 1000 IU vitamin D per day and the increase was significant compared to placebo. The fact that vitamin D may be sufficiently absorbed following a fat-free meal (such as orange juice) may be explained by recent findings on the mechanism by which vitamin D is absorbed. It seems that vitamin D is not only absorbed by simple passive diffusion (by incorporation into the micelle), as cholesterol membrane transporters, such as SR-BI, CD36, or NPC1L1, have been shown to be involved in the absorption. Differences in expression levels and the existence of functional polymorphisms in the genes encoding these proteins may also contribute to the large inter-individual variation in postprandial responses to vitamin D.

Only very few studies are available on the time-plasma concentration profile of vitamin D after intake of an oral dose. Denker et al. studied the pharmacokinetic profile of vitamin D3 after administration of a single D3 dose of either 2800 or 5600 IU, showing that plasma D3 levels increased steadily after the intake and peaked at 9±2.3 h with concentrations returning to near baseline values by 72 h. It is unknown whether the food matrix (including complex formation of vitamin D by encapsulation with whey proteins) affects the bioavailability of vitamin D as assessed by the plasma-time concentration profiles and whether this may influence the inter-individual variability in response to vitamin D supplementation.

The importance of calcium intake, and especially calcium intake from milk products and tablets (supplements) has been investigated in a number of studies, showing discrepant results. A Cochrane meta-analysis has suggested an overall beneficial effect of increased calcium intake from milk products and calcium supplements. However, a recent trial has suggested an increase in blood pressure in the hours following intake of 1000 mg of calcium citrate compared with placebo. It has so far not been investigated whether milk intake causes similar effects on indices of cardiovascular health, including blood pressure and arterial stiffness.

AIM The overall aim of the study is to investigate the influence of different food matrices (including complex-formation with whey proteins) on the bioavailability of vitamin D, as assessed by maximum concentration profiles (Cmax) and the time-concentration curve of D3 in plasma and thereby whether the inter-individual variation in the absorption of vitamin D may depend on delivery system.

Co-primary (null-) hypothesis:

* The food matrix by which D3 is delivered does not affect Cmax of D3 as determined 10h post-dosing.
* The absorption profile (time-concentration curve in terms of Area Under the Curve from 0h to 12h [AUC0-12h]) does not differ according to the food matrix by which D3 is delivered.

Secondary (null-)hypotheses

* Compared with vitamin D provided as droplets, the absorption of D3 is not enhanced by delivery through each of the tested food matrices (i.e., increased Cmax).
* Compared with vitamin D added to juice, the absorption of D3 is not enhanced by whey protein complex-bound D3 (i.e., increased Cmax).
* Treatments do not affect plasma levels of parathyroid hormone (PTH) and ionized calcium.
* The variability to vitamin D supplementation in terms of Cmax is lower if vitamin D is complex-bound to whey proteins as compared to the other tested supplementation methods.
* Arterial stiffness as assessed by tonometry is not affected by milk intake.

Explanatory hypotheses In order to allow for further investigations on indices of importance to responses to vitamin D supplementation, data will be collected on body composition, genetic polymorphisms, cholesterol status, and habitual dietary habits.

MATERIALS AND METHODS

STUDY DESIGN The study is performed as a multiple cross-over study using a balanced latin-square design. This design allows for each participant to function as her own control thereby counterbalancing risk of an adverse influence on results of the order of treatment or other factors such as effect of period, as well as inter-individual variations attributable to e.g., genetic variations, body weight etc. By randomization, each participant will be allocated to receive all the five treatment regimes in a pre-specified order with a 10-21 days wash-out period in-between each of the treatment arms.

The treatment sequences are:

Treatment sequence 1: A B E C D

Treatment sequence 2: B C A D E

Treatment sequence 3: C D B E A

Treatment sequence 4: D E C A B

Treatment sequence 5: E A D B C

Treatment sequence 6: D C E B A

Treatment sequence 7: E D A C B

Treatment sequence 8: A E B D C

Treatment sequence 9: B A C E D

Treatment sequence 10: C B D A E

PROCEDURES FOR HANDLING VITAMIN D SUPPLEMENTATION The supplement will be acquired commercially and stored at the Osteoporosis Clinic, Aarhus University Hospital and kept away from other medication and supplementation. Sub-investigator is responsible for correct handling and dispensing of vitamin D supplement, as well as securing that the supplement will only be used as described in the protocol and that the participants are instructed to take it correct.

PROCEDURES FOR RANDOMIZATION Randomization will be done using a computer generate list. Treatments will not be blinded for the investigator. In terms of comparing juice with or without whey proteins bound-complexes, a single-blind design will be applied, as participants will not be told which of the treatments they are receiving. Each treatment sequence will be allocated to the same number of patients - e.g. 3 participants will be in treatment sequence 1, 3 in treatment sequence 2 etc.

POPULATION Thirty participants will be recruited from the general background population by direct mailing using a list of randomly selected individuals living in the area of Aarhus generated by "Research services" at Statens Serum Institut. The study will be performed during wintertime (November-April).

WITHDRAWAL AND DROPOUT Any participant can at any point drop out of the study without any explanation and will not have to go through a final examination. The investigator can withdraw a participant if this seems necessary for the participant's safety. Dropouts and withdrawals will be noted and explained in the CRF.

Withdrawal will happen in case of one of the following criteria is fulfilled:

* Change in vitamin D supplementation
* Ionized calcium ≥1.40 mmol/L
* Disease or new medication that will influence the study
* Serious adverse effects/symptoms that is expected to be caused by vitamin D supplementation Diseases that occur within 7 days of treatments can be a possible cause of participation in the study. Sub-investigator can in this time frame be contacted in order to investigate whether it is a cause of the vitamin D supplementation. In case it is, the symptoms or disease will be followed until it is cured or have become chronic.

EXAMINATIONS Participants will be examined 5 times over a time period of 6 to 12 weeks. At each visit, the participants will arrive fasting before 9am and will stay at the department until blood sampling at 12 hours is taken. Hereafter, the participants is free to go home and come back the following day for the 24 hours blood sampling and delivering the urine samples or stay the night at the hospital. During the 12 hours at the department, the participants will get standardized food.

Basic health information and questionnaires:

Participants will answer questionnaires regarding their general health as well as dietary habits and sun exposure.

Biochemistry:

Blood samples will be collected at different time points (0, 2, 4, 6, 8, 10, 12, and 24 hours).

All measurements will be performed when all material from all 30 participants have been collected in order to avoid variation in results. Blood samples will be stored in a biobank for a maximum of 15 years after the end of the study.

Urine samples:

Urine will be collected in 3 batches at the first day of each dosing i.e., from 0-4 hours, from 4-8 hours and from 8-24 hours.

All measurements will be performed when all material from all 30 participants have been collected.

Bone scans:

Dual-Energy X-ray absorptiometry (DXA) and High-Resolution peripheral Quantitative Computed Tomography (HRpQCT):

DXA scanning with the Hologic QDR Discovery scanner. Bone mineral density (BMD) will be measured in lumbar spine (L1-L4), femoral neck, and the distal forearm. Furthermore, total body composition will be determined, including fat- and lean-tissue mass.

A HRpQCT bone scan of the distal radius and tibia will be performed using an Xtreme CT-scanner (SCANCO Medical AG, Switzerland). This will allow for assessment of volumetric BMD for cortical and trabecular bone, bone structure and geometry (including cortical and trabecular thickness, trabecular separation etc.) and bone strength.

Blood pressure measurements and tonometry:

Blood pressure and measurements of arterial stiffness (tonometry) are performed twice in each participant in relation to treatment regimes "C" and "D".

On both occasions, measurements are performed in the morning with the participant in the fasting state. After the measurements are performed, the participant will be provided the intervention together with a breakfast meal. After this, the participant will be fasting until next measurement is performed four hours later.

Office blood pressure (BP) is measured in a sitting position after 5 minutes of rest on the right upper arm using a digital automatic BP monitor. Three BP readings will be performed with 2 minutes of rest in-between. The average of the last two measurements is recorded.

Arterial stiffness and pulse wave velocity (PWV) will be assessed by tonometry using the SphygmoCor system (Xcel; AtCor Medical, Sydney, NSW, Australia). For measurements of carotid-to-femoral PWV, an inflated femoral cuff placed on the right upper thigh combined with carotid applanation tonometry will be used. Measurements are performed in a quiet room. The participant will be resting for 10 minutes in a supine position prior to test start. Brachial BP is measured on the right upper arm and two consecutive BP readings are performed. If BP readings do not differ by > 5 mmHg, the last one is recorded. If BP readings differ by > 5 mmHg, four BP readings are obtained. The average of the last two measurements is recorded. AIx is assessed as the ratio of wave reflection amplitude to central pulse pressure. The mean of two measurements are used in the analyses. Carotid-femoral PWV is assessed as the distance travelled divided by the transit time using the direct carotid-to-cuff distance as measured with a non-stretchable tape (infantometer). A minimum of two measurements is performed. If measurements differs < 0.5 m/s the average of the two measurements is used for analyses. If PWV differs by > 0.5 m/s a third measurement is obtained and the median value is used for analyses. According to general recommendations, the direct carotid-to-cuff distance mean PWV is multiple with 0.8.

PERSPECTIVES The study will provide insight into the bioavailability of vitamin D3 supplementation, including sources of variation. Since Denmark is a country with low latitude and high prevalence of vitamin D insufficiency and fortification of food items is not common or legislated, this study may lead to way to fortifying food items in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Caucasian
* Total plasma 25-hydroxy vitamin D < 50 nmol/L
* Understand oral and written Danish
* Able to consent

Exclusion Criteria:

* Known allergic reaction/intolerance to Vitamin D supplementation / milk products / juice
* Known chronic kidney disease (creatinine > 90 µmol/L), previous kidney transplantation or known kidney artery stenosis
* Known liver disease
* Known gastrointestinal malabsorption
* Current malignant disease
* Hypercalcemia (ionised calcium ≥ 1.33 mmol/L)
* Treatment with diuretics, lithium or current use of steroids
* Current use of calcium and/or vitamin D supplementation
* Planned travel during the intervention period to areas where sun exposure is expected
* Use of solarium
* Treatment with beta-blockers
* Overt cardiovascular disease such as known severe heart failure (NYHA III-IV), previous major heart surgery, pacemaker, arrhythmias (e.g. atrial fibrillations or flutter, second- and third-degree atrioventricular block)

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Cmax of vitamin D3 | 10 hours
  Maximum observed concentration of vitamin D3
AUC of vitamin D3 | 12 hours
  Area under the curve for time-concentration relationships during the absorption phase

SECONDARY OUTCOMES:
Concentration of vitamin D metabolites | 24 hours
  Plasma levels of vitamin D2+D3, 25OHD, 1,25(OH)2D, 24,25(OH)2D and VDBP
Concentration of PTH | 24 hours
  Changes in plasma PTH in response to treatment
Plasma concentration of ion-calcium | 24 hours
  Changes in plasma ionized calcium in response to treatment
Urine concentration of calcium | 24 hours
  Changes in urine calcium in response to treatment
Urine concentration of creatinine | 24 hours
  Changes in urine creatinine in response to treatment
Urine concentration of phosphate | 24 hours
  Changes in urine phosphate in response to treatment
Urine concentration of magnesium | 24 hours
  Changes in urine magnesium in response to treatment
Urine concentration of sodium | 24 hours
  Changes in urine sodium in response to treatment
Urine concentration of potassium | 24 hours
  Changes in urine potassium in response to treatment
Urine osmolality | 24 hours
  Changes in urine osmolality in response to treatment
Systolic and diastolic blood pressure | 4 hours
  Office blood pressure of the upper right arm
Pulse wave velocity | 4 hours
  Assessed by tonometry using SphygmoCor system
Arterial stiffness | 4 hours
  Assessed by tonometry using SphygmoCor system system (Xcel; AtCor Medical, Sydney, NSW, Australia)

OTHER OUTCOMES:
Body composition | Week 4
  Assessed by DXA
Areal BMD | Week 4
  BMD at the lumbar spine, femoral neck and distal forearm assessed by DXA
Bone geometry | Week 4
  Assessed by HRpQCT of distal tibia and distal radius
Volumetric BMD | Week 4
  Assessed by HRpQCT of distal tibia and distal radius
Estimated bone strength | Week 4
  Assessed by HRpQCT of distal tibia and distal radius
Plasma concentrations of bone turnover markers | Week 4
  Plasma levels of bone-specific alkaline phosphatase, osteocalcin, procollagen type I N-terminal propeptide (P1NP), C-terminal telopeptide (CTX), sclerostin and fibroblast growth factor 23 (FGF-23)
Exome sequencing | 24 hours
  Genetic variants of importance to vitamin D metabolism
Plasma concentrations of total cholesterol, triglycerides, LDL- and HDL-cholesterol | 24 hours
  Cholesterol status
Plasma concentrations of metabolites | 24 hours
  Metabolomics analyses: Blood samples for nuclear magnetic resonance and liquid chromatography mass spectrometry analyses
General health | Week 1
  Questionnaire
Dietary habits | Week 1
  Questionnaire
Sun exposure | Week 1
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rejnmark, Principal Investigator — Dept. of Endocrinology and Internal Medince, The Osteoporosis Clinic
Locations (1):
- Dept. of Endocrinology and Internal Medicine, The Osteoporosis Clinic, Aarhus N, Denmark

REFERENCES:
- [Background] Pedersen JN, Frislev HS, Pedersen JS, Otzen DE. Using protein-fatty acid complexes to improve vitamin D stability. J Dairy Sci. 2016 Oct;99(10):7755-7767. doi: 10.3168/jds.2016-11343. Epub 2016 Jul 27. PMID 27474981
- [Background] Bouillon R, Carmeliet G, Daci E, Segaert S, Verstuyf A. Vitamin D metabolism and action. Osteoporos Int. 1998;8 Suppl 2:S13-9. doi: 10.1007/pl00022727. No abstract available. PMID 10197177
- [Background] Heaney RP, Davies KM, Chen TC, Holick MF, Barger-Lux MJ. Human serum 25-hydroxycholecalciferol response to extended oral dosing with cholecalciferol. Am J Clin Nutr. 2003 Jan;77(1):204-10. doi: 10.1093/ajcn/77.1.204. PMID 12499343
- [Background] Shab-Bidar S, Bours S, Geusens PP, Kessels AG, van den Bergh JP. Serum 25(OH)D response to vitamin D3 supplementation: a meta-regression analysis. Nutrition. 2014 Sep;30(9):975-85. doi: 10.1016/j.nut.2013.12.020. Epub 2014 Jan 10. PMID 24993750
- [Background] Shab-Bidar S, Bours SP, Geusens PP, van der Velde RY, Janssen MJ, van den Bergh JP. Suboptimal effect of different vitamin D3 supplementations and doses adapted to baseline serum 25(OH)D on achieved 25(OH)D levels in patients with a recent fracture: a prospective observational study. Eur J Endocrinol. 2013 Oct 1;169(5):597-604. doi: 10.1530/EJE-13-0068. Print 2013 Nov. PMID 23959785
- [Background] Binkley N, Borchardt G, Siglinsky E, Krueger D. DOES VITAMIN D METABOLITE MEASUREMENT HELP PREDICT 25(OH)D CHANGE FOLLOWING VITAMIN D SUPPLEMENTATION? Endocr Pract. 2017 Apr 2;23(4):432-441. doi: 10.4158/EP161517.OR. Epub 2017 Jan 17. PMID 28095046
- [Background] Tanner JT, Smith J, Defibaugh P, Angyal G, Villalobos M, Bueno MP, McGarrahan ET, Wehr HM, Muniz JF, Hollis BW, et al. Survey of vitamin content of fortified milk. J Assoc Off Anal Chem. 1988 May-Jun;71(3):607-10. PMID 3391970
- [Background] Holick MF, Shao Q, Liu WW, Chen TC. The vitamin D content of fortified milk and infant formula. N Engl J Med. 1992 Apr 30;326(18):1178-81. doi: 10.1056/NEJM199204303261802. PMID 1313548
- [Background] Chen TC, Shao A, Heath H 3rd, Holick MF. An update on the vitamin D content of fortified milk from the United States and Canada. N Engl J Med. 1993 Nov 11;329(20):1507. doi: 10.1056/NEJM199311113292021. No abstract available. PMID 8413473
- [Background] Gallagher JC, Sai A, Templin T 2nd, Smith L. Dose response to vitamin D supplementation in postmenopausal women: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):425-37. doi: 10.7326/0003-4819-156-6-201203200-00005. PMID 22431675
- [Background] Nelson ML, Blum JM, Hollis BW, Rosen C, Sullivan SS. Supplements of 20 microg/d cholecalciferol optimized serum 25-hydroxyvitamin D concentrations in 80% of premenopausal women in winter. J Nutr. 2009 Mar;139(3):540-6. doi: 10.3945/jn.108.096180. Epub 2009 Jan 21. PMID 19158226
- [Background] Blum M, Dallal GE, Dawson-Hughes B. Body size and serum 25 hydroxy vitamin D response to oral supplements in healthy older adults. J Am Coll Nutr. 2008 Apr;27(2):274-9. doi: 10.1080/07315724.2008.10719700. PMID 18689559
- [Background] Wagner D, Hanwell HE, Schnabl K, Yazdanpanah M, Kimball S, Fu L, Sidhom G, Rousseau D, Cole DE, Vieth R. The ratio of serum 24,25-dihydroxyvitamin D(3) to 25-hydroxyvitamin D(3) is predictive of 25-hydroxyvitamin D(3) response to vitamin D(3) supplementation. J Steroid Biochem Mol Biol. 2011 Sep;126(3-5):72-7. doi: 10.1016/j.jsbmb.2011.05.003. Epub 2011 May 13. PMID 21605672
- [Background] Fu L, Yun F, Oczak M, Wong BY, Vieth R, Cole DE. Common genetic variants of the vitamin D binding protein (DBP) predict differences in response of serum 25-hydroxyvitamin D [25(OH)D] to vitamin D supplementation. Clin Biochem. 2009 Jul;42(10-11):1174-7. doi: 10.1016/j.clinbiochem.2009.03.008. Epub 2009 Mar 18. PMID 19302999
- [Background] Zhao LJ, Zhou Y, Bu F, Travers-Gustafson D, Ye A, Xu X, Hamm L, Gorsage DM, Fang X, Deng HW, Recker RR, Lappe JM. Factors predicting vitamin D response variation in non-Hispanic white postmenopausal women. J Clin Endocrinol Metab. 2012 Aug;97(8):2699-705. doi: 10.1210/jc.2011-3401. Epub 2012 May 14. PMID 22585090
- [Background] Borel P, Caillaud D, Cano NJ. Vitamin D bioavailability: state of the art. Crit Rev Food Sci Nutr. 2015;55(9):1193-205. doi: 10.1080/10408398.2012.688897. PMID 24915331
- [Background] Reboul E. Intestinal absorption of vitamin D: from the meal to the enterocyte. Food Funct. 2015 Feb;6(2):356-62. doi: 10.1039/c4fo00579a. PMID 25367187
- [Background] Thompson GR, Lewis B, Booth CC. Absorption of vitamin D3-3H in control subjects and patients with intestinal malabsorption. J Clin Invest. 1966 Jan;45(1):94-102. doi: 10.1172/JCI105327. No abstract available. PMID 4285212
- [Background] Iqbal J, Hussain MM. Intestinal lipid absorption. Am J Physiol Endocrinol Metab. 2009 Jun;296(6):E1183-94. doi: 10.1152/ajpendo.90899.2008. Epub 2009 Jan 21. PMID 19158321
- [Background] Raimundo FV, Lang MA, Scopel L, Marcondes NA, Araujo MG, Faulhaber GA, Furlanetto TW. Effect of fat on serum 25-hydroxyvitamin D levels after a single oral dose of vitamin D in young healthy adults: a double-blind randomized placebo-controlled study. Eur J Nutr. 2015 Apr;54(3):391-6. doi: 10.1007/s00394-014-0718-8. Epub 2014 May 23. PMID 24853643
- [Background] Tangpricha V, Koutkia P, Rieke SM, Chen TC, Perez AA, Holick MF. Fortification of orange juice with vitamin D: a novel approach for enhancing vitamin D nutritional health. Am J Clin Nutr. 2003 Jun;77(6):1478-83. doi: 10.1093/ajcn/77.6.1478. PMID 12791627
- [Background] Biancuzzo RM, Young A, Bibuld D, Cai MH, Winter MR, Klein EK, Ameri A, Reitz R, Salameh W, Chen TC, Holick MF. Fortification of orange juice with vitamin D(2) or vitamin D(3) is as effective as an oral supplement in maintaining vitamin D status in adults. Am J Clin Nutr. 2010 Jun;91(6):1621-6. doi: 10.3945/ajcn.2009.27972. Epub 2010 Apr 28. PMID 20427729
- [Background] Reboul E, Goncalves A, Comera C, Bott R, Nowicki M, Landrier JF, Jourdheuil-Rahmani D, Dufour C, Collet X, Borel P. Vitamin D intestinal absorption is not a simple passive diffusion: evidences for involvement of cholesterol transporters. Mol Nutr Food Res. 2011 May;55(5):691-702. doi: 10.1002/mnfr.201000553. Epub 2011 Jan 31. PMID 21280209
- [Background] Masson CJ, Plat J, Mensink RP, Namiot A, Kisielewski W, Namiot Z, Fullekrug J, Ehehalt R, Glatz JF, Pelsers MM. Fatty acid- and cholesterol transporter protein expression along the human intestinal tract. PLoS One. 2010 Apr 29;5(4):e10380. doi: 10.1371/journal.pone.0010380. PMID 20454462
- [Background] Desmarchelier C, Borel P, Goncalves A, Kopec R, Nowicki M, Morange S, Lesavre N, Portugal H, Reboul E. A Combination of Single-Nucleotide Polymorphisms Is Associated with Interindividual Variability in Cholecalciferol Bioavailability in Healthy Men. J Nutr. 2016 Dec;146(12):2421-2428. doi: 10.3945/jn.116.237115. Epub 2016 Oct 26. PMID 27798339
- [Background] Denker AE, Lazarus N, Porras A, Ramakrishnan R, Constanzer M, Scott BB, Chavez-Eng C, Woolf E, Maganti L, Larson P, Gottesdiener K, Wagner JA. Bioavailability of alendronate and vitamin D(3) in an alendronate/vitamin D(3) combination tablet. J Clin Pharmacol. 2011 Oct;51(10):1439-48. doi: 10.1177/0091270010382010. Epub 2010 Dec 8. PMID 21148044
- [Background] Kazmi SA, Vieth R, Rousseau D. Vitamin D3 fortification and quantification in processed dairy products. International Dairy Journal 17:753-759, 2007
- [Background] Cormick G, Ciapponi A, Cafferata ML, Belizan JM. Calcium supplementation for prevention of primary hypertension. Cochrane Database Syst Rev. 2015 Jun 30;2015(6):CD010037. doi: 10.1002/14651858.CD010037.pub2. PMID 26126003
- [Background] Billington EO, Bristow SM, Gamble GD, de Kwant JA, Stewart A, Mihov BV, Horne AM, Reid IR. Acute effects of calcium supplements on blood pressure: randomised, crossover trial in postmenopausal women. Osteoporos Int. 2017 Jan;28(1):119-125. doi: 10.1007/s00198-016-3744-y. Epub 2016 Aug 20. PMID 27543500
- [Background] Van Bortel LM, Laurent S, Boutouyrie P, Chowienczyk P, Cruickshank JK, De Backer T, Filipovsky J, Huybrechts S, Mattace-Raso FU, Protogerou AD, Schillaci G, Segers P, Vermeersch S, Weber T; Artery Society; European Society of Hypertension Working Group on Vascular Structure and Function; European Network for Noninvasive Investigation of Large Arteries. Expert consensus document on the measurement of aortic stiffness in daily practice using carotid-femoral pulse wave velocity. J Hypertens. 2012 Mar;30(3):445-8. doi: 10.1097/HJH.0b013e32834fa8b0. PMID 22278144